CLINICAL TRIAL: NCT00972985
Title: Acute Effect of Three Neuroactive Drugs on Brain Activity Measured by MEG, EEG and the Synchronous Neural Interaction Test
Brief Title: Acute Effect of Three Neuroactive Drugs Measured by Magnetoencephalography (MEG), Electroencephalography (EEG) and the Synchronous Neural Interaction Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orasi Medical, Inc. (Industry)
Responsible Party: Todd Verdoorn, Ph.D., Chief Scientific Officer, Orasi Medical, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ADE 09-01
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Healthy Control subjects
MeSH Terms: interventions — Modafinil; Methylphenidate; Lorazepam; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- modafinil (Experimental): All healthy control subjects receive modafinil in this crossover design
  Interventions: Drug: modafinil
- methylphenidate (Experimental): All healthy control subjects receive methylphenidate in this crossover design
  Interventions: Drug: methylphenidate
- lorazepam (Experimental): All healthy control subjects receive lorazepam in this crossover design
  Interventions: Drug: lorazepam
- placebo (Placebo Comparator): All healthy control subjects receive placebo in this crossover design
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: modafinil — oral tablet, 100 mg, single acute dose
  Other Names: Provigil
  Arms: modafinil
Drug: methylphenidate — oral tablet, 20 mg, single acute dose
  Other Names: Ritalin
  Arms: methylphenidate
Drug: lorazepam — oral tablet, 1 mg, single, acute dose
  Other Names: Ativan
  Arms: lorazepam
Drug: placebo — oral tablet, single acute dose
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
This placebo-controlled crossover study is intended to measure the effect of three, common neuroactive medications on brain activity measured by magnetoencephalography (MEG) and electroencephalography (EEG). This study will conduct MEG and EEG scans as well as simple cognition testing on 15 healthy volunteers over 4 study days. Subjects will receive placebo on one of the study days, and either 100 mg modafinil p.o., 20 mg methylphenidate p.o., or 1 mg lorazepam p.o. on remaining study days. Medication administration will be randomized according to study day so that each subject will receive the medications in random order. Brain activity will be measured by MEG and EEG in each subject a total of 4 times each study day: prior to medication administration and 2, 4, and 6 hours after medication administration. Cognition testing will be performed at pre-medication baseline and immediately after each post-medication scan time. This study will test the hypothesis that changes in brain functional activity can be accurately measured in healthy volunteer subjects after single, acute doses of modafinil, methylphenidate and lorazepam.

DETAILED DESCRIPTION:
This study uses a placebo-controlled, crossover design to investigate the effect of modafinil (100 mg, p.o.), methylphenidate (20 mg, p.o.), and lorazepam (1 mg, p.o.) in 15 healthy male volunteers. The acute effect of the medications will be measured by MEG, EEG and simple cognition testing. Study procedures will be performed over 5 separate days. During an initial screening visit, Study Day 1, subjects will consent to enroll and undergo clinical evaluation sufficient to determine they are eligible to participate in the study. Upon qualification and enrollment, subjects will be randomly assigned to receive either placebo or one of the active medications on Study Days 2 - 5. Medications or placebo will be administered orally. Subjects will arrive at the MEG center in the morning on Study Day 2 and baseline MEG and EEG scans will be performed along with baseline cognition testing. The medication or placebo will be administered immediately following the baseline scans and cognition testing. Additional MEG and EEG scans will be conducted 2, 4, and 6 hours after medication or placebo administration. On Study Days 3 - 5, subjects will undergo identical procedures but will be crossed over to receive the alternate medication or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male between 18 and 35 years of age at the time of screening.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is a non-smoker.
* Subject is judged to be in good health based on medical history and brief physical examination.
* Subject has normal or corrected to normal visual and auditory acuity.
* Subject agrees to refrain from caffeine 24 hours prior to and then throughout each Study Day.
* Subject agrees to refrain from using alcohol for 48 hours prior to and then throughout each Study Day.

Exclusion Criteria:

* Subject has a diagnosis of a significant neurological condition including Alzheimer's disease, Parkinson's disease, vascular dementia, Lewy body dementia or frontal temporal dementia, human immunodeficiency virus, multiple sclerosis, or severe traumatic brain injury.
* Subject has a history of primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, delusional disorder) or bipolar disorder.
* Subject has a history of seizures, epilepsy, stroke, peripheral neuropathy, head trauma with persistent post-concussive symptoms, ADHD, dyslexia or other clinically significant neurological disease or cognitive impairment.
* Subject has a lifetime or current history of alcohol or substance abuse/dependence.
* Subject has a history of multiple or severe allergies, or has had an anaphylactic reaction or intolerability to prescription or non-prescription drugs or food. This includes a documented or subject-verified allergy.
* Subject had an MRI 2 weeks prior to Study Day 2.
* Subject has metal braces or pacemaker that may interfere with the MEG scan.
* Subject is unable to complete the MEG scan procedure.
* The investigator has any concern regarding the safe participation of a subject in the study, or if for any other reason the investigator considers the subject inappropriate for study participation.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study will be identification and characterization of a pattern of synchronous brain activity that is specifically altered by administration of active medications compared to pre-medication baseline and placebo. | The study will require 5 days for each subject. Data collection for the study is expected to require approximately 12 weeks.

SECONDARY OUTCOMES:
Standard frequency-domain analysis of the MEG data to identify and quantify medication-induced changes in signal power in particular frequency bands associated with brain functional activity | Data collection for the study is expected to require approximately 12 weeks.
Standard frequency-domain and time-domain analysis of EEG data to generate direct comparisons between MEG and EEG results; | Data collection for the study is expected to require approximately 12 weeks.
Orasi will apply its data analysis technology to the EEG data in an effort to compare the time-domain correlations measured by EEG to those measured with MEG; | Data collection for the study is expected to require approximately 12 weeks.
Orasi will compare the pattern of cross-correlations observed with medications to those observed in our database of healthy and disease subjects; | Data collection for the study is expected to require approximately 12 weeks.
The results of standard cognitive tests designed to identify the known effects of medications. | Data collection for the study is expected to require approximately 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Concetta Forchetti, MD, PhD, Principal Investigator — Alexian Brothers Neuroscience Institute
Locations (1):
- Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois, United States